CLINICAL TRIAL: NCT06025981
Title: Clinical Study of the Effects of a Robotic Walker and Immersive Technology for Hip Fracture Rehabilitation in the Elderly
Brief Title: Clinical Study of the Effects of a SWalker II and VR for Hip Fracture Rehabilitation in the Elderly
Acronym: SWalker-VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Werium Assistive Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SWalker-II-VR
Record Dates: First submitted 2023-06-20; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-07

CONDITIONS: Hip Fractures; Gait Disorders in Old Age
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: The model is that of a prospective, longitudinal, multicenter, randomized controlled trial (RCT), open-label and analytical:
  * RCT: A rehabilitation intervention with SWalker (experimental group) and a conventional one (control group) will be implemented, following randomization.
  * Prospective longitudinal: Study requiring follow-up of patients during the hip fracture rehabilitation period.
  * Open multicenter: Inclusion is not limited to any individual who meet the inclusion criteria from Valle de la Oliva-Majadahonda, Ciempozuelos, Mirasierra and Moratalaz nursing homes.
  * Analytical: Results are presented in a descriptive way and entering into the analytical statistics of comparison and relationship. analytical comparison and relationship.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preliminary Phase (Other): 20 healthy subjects will perform an experimental session for characterization of functional status with clinical scales; characterization of gait with SWalker using ROM and EMG at different speeds and weight bearing; and assessment of system usability with VR using standardized questionnaires.
  Interventions: Other: Preliminary Phase
- Phase I and II (Other): In both phases 100 subjects will perform a gait rehabilitation intervention program (phase 1) and maintenance (phase 2), in which they will employ the use of the robotic walker and virtual reality depending on the group and phase. The evolution of functional clinical parameters will be studied for both groups and phases.
  Interventions: Other: Phase I - Early gait rehabilitation; Other: Phase II - Maintenance gait function ( with VR)

INTERVENTIONS:
Other: Preliminary Phase — In the preliminary phase, the characterization of the functionality of the SWalker robotic system, as well as the functionality of the Virtual Reality system, will be carried out. All descriptive usability questionnaires completed by the participants and electro-biomechanical parameters will be collected using the robot's measurement systems to analyze the functionality.
  Arms: Preliminary Phase
Other: Phase I - Early gait rehabilitation — In the first phase, the participants will carry out the rehabilitation program for hip fracture in acute phase that will last 6 weeks. Participants will be randomized between control and experimental groups. In which the therapeutic intervention is based on the usual rehabilitation guidelines that integrate exercises aimed at improving strength, gait, functional mobility and balance. In the case of the experimental group, a robotic walker will be used to practice walking.
  Arms: Phase I and II
Other: Phase II - Maintenance gait function ( with VR) — In the second phase, participants will carry out a 6-week program to consolidate walking function. Participants will be randomized between control and experimental groups. In which the therapeutic intervention is based on the use of the robotic system for gait exercise. In the case of the experimental group, the use of virtual reality will also be integrated.
  Arms: Phase I and II

SUMMARY:
This project is structured in two distinct phases. The first phase deals with the recovery of the hip fracture in the acute phase up to ambulation, and the second is understood as the continuation of functional improvement of gait. In the first phase, the aim is to evaluate the effects of the use of the robotic device (SWalker) on the physical improvement of the patient. While in the second phase, the objective is to evaluate the effects of virtual reality technology combined with the use of the SWalker.Therefore, the following specific objectives are identified:

* Phase I: To analyze the effects of SWalker application in patients with acute hip fracture on clinical parameters of rehabilitation.
* Phase II: To study the effects of the application of the SWalker combined with immersive technology in people with impaired gait function after hip fracture.

DETAILED DESCRIPTION:
In the preliminary phase, the usability and acceptance of the SWalker II system combined with virtual reality is evaluated with a group of healthy subjects. For this purpose, an exposure session and the evaluation of the system based on questionnaires are carried out. On the other hand, a gait characterization session (capture of ROM and EMG) is performed inside and outside the walker with different speeds and weight loads.

In the first phase of the clinical study, patients with hip fractures in the early rehabilitation phase were recruited. They are randomly assigned to a control group or experiment group. And for a period of 6 weeks, both groups carry out the same rehabilitation exercise program based on strength, balance and ambulation exercise. The difference is that the experimental group performs the rehabilitation exercises with the SWalker, and the control group performs these exercises with conventional parallel bars.

In the second phase of the clinical study, these same patients who have passed the first pass, move on to a 6-weeks program of maintenance and improvement of gait function. Again, they are divided into 2 groups, control and experimental. So the control group will perform walking exercises with the Swalker and conventional balance exercises and the experimental group will perform walking and balance exercises with SWalker and virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes over 65 years of age,
* Patients with a height of less than 180 cm,
* Patients weighing less than 90 kg,
* Patients who have suffered a hip fracture* and wish to participate in the study.
* In addition, they must sign and understand the informed consent form.

Exclusion Criteria:

* Cognitive status insufficient to understand and execute instructions given by the physiotherapist.

  * Patients needing rehabilitation after hip fracture may vary from a few days to a few weeks after the period of occurrence of the hip fracture, depending on the complications that could arise and the type of surgery used, with a pre-set limit of one month.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Pain | 6 weeks
  The evolution of the functional clinical scales will be studied (pain): Pain by means of the Verbal Rating Scale, a five-point scale and consists of a list of adjectives describing various levels of symptom intensity (0= no itch, 1= mild itch, 2= moderate itch , 3= severe itch and 4=very severe itch).
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Autonomy/independence. Ambulation | 6 weeks
  The evolution of the functional clinical scales will be studied (autonomy/independence): Functional limitation in early post-acute phase by means of Cumulative Ambulation Score (CAS) (Physical test). The CAS describes the patient's independence with regard to three activities (getting in and out of bed, sit-to-stand-to-sit from a chair, and walking). Each activity is assessed on a three-point ordinal scale from 0-2 (0 = Not able to, despite human assistance and verbal cueing, 1 = Able to, with human assistance and/or verbal cueing from one or more persons, 2 = Able to safely, without human assistance or verbal cueing, use of a walking aid allowed) resulting in a total daily CAS score ranging from 0 to 6.
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Strength | 6 weeks
  The evolution of the functional clinical scales will be studied (strength): Muscle strength of the lower limbs through quadriceps extension test or lower limb dynamometer (physiological parameter).
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Gait | 6 weeks
  The evolution of the functional clinical scales will be studied (gait and balance): Gait speed using the 10 metre Walk Test (10MWT) (physical test), provided the patient can walk without human assistance; The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. The total time is recorded in m/s. Household Ambulator <0.40 m/s; Limited Community Ambulator 0.40 to <0.80 m/s; Community Ambulator ≥0.80 m/s.
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Autonomy/independence. Fear of falling | 6 weeks
  The evolution of the functional clinical scales will be studied (autonomy/independence): Fear of falling by means of the Falls Efficacy Scale International (questionnaire); The total score ranges from 16 to 64, where 16 indicates "no concern" and 64 indicates "extremely concerned about falling" during the performance of the specific activities suggested by the questionnaire.
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Autonomy/independence. Quality of life. | 6 weeks
  The evolution of the functional clinical scales will be studied (autonomy/independence): Quality of life through the 36-Item Short Form Survey (SF-36) (questionnaire). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Autonomy/independence. Mobility | 6 weeks
  The evolution of the functional clinical scales will be studied (autonomy/independence): Mobility using the New Mobility Test (Physical test), also known as Parker Mobility Test. It is a composite score of the patient's ability to perform: indoor walking, outdoor walking, and shopping, providing a score between 0 and 3 (0 - not at all, 1 - with help from another person, 2 - with an aid, 3 - no difficulty) for each function, resulting in a total score from 0 (no walking ability at all) to 9 (fully independent) .
Effects of robotic system (SWalker + VR) use in gait rehabilitation - Gait and Balance | 6 weeks
  The evolution of the functional clinical scales will be studied (gait and balance): Functionality through the Timed Up & Go test (physical test). Its score is the time spent (seconds) while the subject is standing from an armchair, walking 3 meters, returning to the chair walking 3 additional meters and sitting down. It is considered that scores of 10 seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance.

SECONDARY OUTCOMES:
Usability of virtual reality system combined with the robotic system (SWalker) - Presence | 1 week
  Descriptive analysis of system's usability: questionnaires will be collected to assess the following aspects: feeling of presence in the virtual environment using the Presence Questionnaire, PQ); Presence Questionnaire consists of 32 questions each on a 1 to 7 scale. The final presence score is the sum of 32 such questions. A total score < 4 is considered unsatisfactory, and score >4 is considered satisfactory.
Usability of virtual reality system combined with the robotic system (SWalker) - Safety | 1 week
  Descriptive analysis of system's safety: the Simulator Sickness Questionnaire, SSQ, will be collected to assess the presence of adverse effects due to cybersickness. Each item is rated with the scale from none (0), slight (1), moderate (2) to severe (3). Through some calculations, four representative scores can be found. Nausea-related subscore (N), Oculomotorrelated subscore (O), Disorientation-related subscore (D) are the scores for the symptoms for the specific aspects. Total Score (TS) is the score representing the overall severity of cybersickness experienced by the users of virtual reality systems. It is suggested that total scores can be associated with negligible (< 5), minimal (5 - 10), significant (10 - 15), and concerning (15 - 20) symptoms. A simulator resulting in total scores above 20 is considered "bad".
Feasibility of robotic system (SWalker) - Gait | 1 week
  Gait and balance using the SWalker will be studied in a 4-meter walk at 3 different speeds for 0%, 25% and 50% of weight bearing: Timed Up & Go test (physical test). Its score is the time spent (seconds) while the subject is standing from an armchair, walking 3 meters, returning to the chair walking 3 additional meters and sitting down. It is considered that scores of 10 seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance.
Feasibility of robotic system (SWalker) - Hip ROM | 1 week
  Hip range of motion (ROM) (physiological parameter) will be studied (using the SWalker) in a 4-meter walk at 3 different speeds for 0%, 25% and 50% of weight bearing. In general, the average range of motion for hip extension in a healthy person is about 20-30 degrees out of a neutral stance.
Usability of virtual reality system combined with the robotic system (SWalker) - Usability | 1 week
  Descriptive analysis of system's usability: questionnaires will be collected to assess the following aspects: general usability of the system using the System Usability Scale (questionnaire) and the Post-Study System Usability Questionnaire. The System Usability Scale score ranges from 0 to 100, being a total score above 80.3 considered excellent, a score between 68 - 80.3 is considered good, and below 68 is considered poor. The Post-Study System Usability Questionnaire score starts with 1 (strongly agree) and ends with 7 (strongly disagree). The lower the score, the better the performance and satisfaction, considering 4 neutral score.
Feasibility of robotic system (SWalker) - Gait and Balance | 1 week
  Gait and balance using the SWalker will be studied in a 4-meter walk at 3 different speeds for 0%, 25% and 50% of weight bearing: the 10-meter walking speed (10MWT) (physical test). The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. The total time is recorded in m/s. Household Ambulator <0.40 m/s; Limited Community Ambulator 0.40 to <0.80 m/s; Community Ambulator ≥0.80 m/s.
Feasibility of robotic system (SWalker) - Physical Performance | 1 week
  Gait and balance using the SWalker will be studied in a 4-meter walk at 3 different speeds for 0%, 25% and 50% of weight bearing: the Short Physical Performance Battery test (SPPB) (physical test). SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with possible sarcopenia but no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness. Persons with a score of 2 or lower who have sarcopenia, and mobility disability are determined to be disabled.
Feasibility of robotic system (SWalker) - EMG activity | 1 week
  The electromyographic (EMG) activity of the two leg muscles (Tibialis anterior [TA] and Soleus [SOL]) (physiological parameter) will be studied (using the SWalker) in a 4-meter walk at 3 different speeds for 0%, 25% and 50% of weight bearing. It will be studied the peak amplitudes (mV) for left and right leg muscles s-EMG activity.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Werium Assistive Solutions, Arganda, Madrid
  - Albertia Servicios Sociosanitarios, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa V, Rojo A, Lopez-Lopez S, Pareja-Galeano H, Velasquez A, Perea L, Raya R. Evaluating the Usability and Safety of Virtual Reality Application Combined with the SWalker for Functional Gait Rehabilitation. Games Health J. 2024 Oct;13(5):397-405. doi: 10.1089/g4h.2023.0172. Epub 2024 May 17. PMID 38757664